CLINICAL TRIAL: NCT04723173
Title: Quality Control of CE-Certified Phonak Hearing Aids - 2020_43
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sonova AG (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Other
Other Study IDs: Sonova2020_43
Record Dates: First submitted 2021-01-22; First posted 2021-01-25 (Actual); Results first posted 2022-02-17 (Actual); Last update posted 2022-03-11 (Actual); Status verified 2021-08

CONDITIONS: Hearing Loss
MeSH Terms: conditions — Hearing Loss

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental device: Noise reduction on (Experimental): The noise reduction is activated. The feature shall support the hearing aid user in noisy situation and shall reduce the listening effort in these special situations.
  Interventions: Device: Feature for noise reduction (on)
- Experimental device: Noise reduction off (Active Comparator): To compare the advantage of the special noise reduction feature the tests will be done additionally with the deactivated feature.
  Interventions: Device: Feature for noise reduction (off)

INTERVENTIONS:
Device: Feature for noise reduction (on) — The noise reduction feature shall support the hearing aid user in noisy situations and shall reduce the listening effort.
  Arms: Experimental device: Noise reduction on
Device: Feature for noise reduction (off) — To show the advantage of the noise reduction feature there is a comparison without the feature necessary.
  Arms: Experimental device: Noise reduction off

SUMMARY:
Phonak Hearing Systems pass through different development and study stages. At an early stage, feasibility studies are conducted to investigate new algorithms, features and functions in an isolated manner. If the benefit is proven, their performance is then investigated regarding interdependency between all available algorithms, features and functions running in parallel in a hearing aid (pivotal/pre-validation studies) and, as a result, they get optimized. Afterwards, and prior to product launch, the Phonak Hearing Systems undergo a final quality control in terms of clinical trials. This is a pre-validation study, investigating optimized algorithms, features, functions and wearing comfort. This will be a clinical investigation which will be conducted mono centric at Sonova AG Headquarters based in Stäfa (Switzerland).

DETAILED DESCRIPTION:
The study will compare different features of the Phonak behind the ear device activated and deactivated, for example the noise reduction feature. There shall be differences in listening effort, awareness and sound quality shown. The study shall show the advantages especially for people with severe to profound hearing losses. This will be a clinical investigation which will be conducted mono centric at Sonova AG Headquarters based in Stäfa (Switzerland).

ELIGIBILITY:
Inclusion Criteria:

* Adult hearing impaired persons (minimum age: 18 years, severe to profound Hearing loss)
* Good written and spoken (Swiss) German language skills
* Healthy outer ear
* Ability to fill in a questionnaire (p/eCRF) conscientiously
* willingness to wear Behind-the-ear hearing aids
* Informed Consent as documented by signature

Exclusion Criteria:

* Contraindications to the MD in this study, e.g. known hypersensitivity or allergy to the investigational product
* Limited mobility and not in the position to attend weekly appointments in Stäfa (Switzerland)
* Limited ability to describe listening impressions/experiences and the use of the hearing aid
* Inability to produce a reliable hearing test result
* Known psychological problems

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2020-12-07 (Actual); Primary Completion 2021-05-11 (Actual); Study Completion 2021-06-07 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Sonova AG, Stäfa, Canton of Zurich, Switzerland

RESULTS

PARTICIPANT FLOW:
Groups:
- Study Population: This was a crossover design, in which all participants undertook the same conditions.
  The conditions (different hearing aid settings) were completed in a randomized order during a single study appointment. Therefore the number starting each period will not match the number completing the previous period.
  The study started with 10 participants in total. Single tests (test period 2 and 3) started just with 9 participants, because there was 1 withdrawal. Test period 2 were completed with 1 participant less, than test period 3 started. That was possible, because the tests were independent and 1 participant was not able to perform the test is period 2, but was able to perform the test in period 3.
Period: Measure of Detection Threshold (in dB)
Arm/Group | Study Population
Started | 10
Feature for Soft Sounds On | 10
Feature for Soft Sounds Off | 10
Completed | 10
Not Completed | 0
Period: Subjective Listening Effort Scaling
Arm/Group | Study Population
Started | 9 (The test in this test period is independent (also temporally) from the previous test period. That is the reason, why the number of participants, who started this test period is lesser than the number of participants, who completed the previous period.)
DNC on | 9
DNC Off | 9
Completed (This test compared the activated and deactivated feature for noisy situations. It was done in a single appointment and each participant performed randomized the test with both conditions. The reason for the smaller sample size (10 started the study, just 9 this test period) is that 1 participant left the study prior to the test and 1 participant started the test, but was not able to perform the test as the study protocol required. Nevertheless this participant completed the rest of the study.) | 8
Not Completed | 1
Not completed — One participant was not able to perform the test as required by the study protocol. | 1
Period: Subjective Ratings of Sound Samples
Arm/Group | Study Population
Started | 9 (The test in this test period is independent (also temporal) from the previous test period. That is the reason, why the number of participants, who started this test period is greater than the number of participants, who completed the previous period.)
DNC on | 9
DNC Off | 9
Completed | 9 (All participants completed this study period, but just the results of 8 participants could be used. This was because technical issues limited the reliability of the measures made for one participant. N.B. this test was independent from the other tests in the study. Therefore the results are not influenced by other test periods. The number of people included in the analysis described here relates only to this test.)
Not Completed | 0

BASELINE CHARACTERISTICS:
Groups:
- Study Population: This was a crossover design, in which all participants undertook the same conditions.
Arm/Group | Study Population
Number analyzed (Participants) | 10
Age, Continuous [Mean (Full Range); unit: years] | 62.7 [49 to 75]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4
  Male | 6
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  Switzerland | 10

OUTCOME MEASURES:

1. Primary Outcome: Subjective Listening Effort Scaling
Description: A listening effort scaling procedure ('ACALES'; Krueger et al, 2017) was performed with noise cancellation on and off.
  ACALES is adaptive, altering the signal-to-noise ratio (SNR) at which speech is presented. Therefore it is not a simple rating scale.
  For each stimulus, a rating (14-point scale ranging from 1='effortless' to 14= 'only noise') was given for how "effortful" it was following speech.
  This results in 2-D data: a list of presentation SNRs (different for each participant), and respective participant ratings.
  Given the format of this data, it cannot be summarized using standard descriptive statistics.
  We defined SNR as the dependent variable and fitted a linear mixed effects model, with the predictors: listening effort rating & intervention (treating participants as a random factor), characterizing SNR over the entire rating scale.
  The values reported represent the estimated marginal means of SNR for each intervention, averaged across effort ratings & participants.
Time Frame: 2 weeks
Population: In total there were 8 participants, who performed this test. It was a crossover- design, so each participant completed both arms during a single appointment in a randomized order.
  9 participants started the test, but 1 was not able to perform the test, so the procedure was stopped for this participant and no data was collected.
Measure: Mean (95% Confidence Interval); unit: SNR (dB)
Groups:
- Noise Reduction on: The noise reduction is activated. The feature shall support the hearing aid user in noisy situations and shall reduce the listening effort in these special situations.
  Feature for noise reduction (on): The noise reduction feature shall support the hearing aid user in noisy situations and shall reduce the listening effort.
  Feature for noise reduction (off): To show the advantage of the noise reduction feature there is a comparison without the feature necessary.
- Noise Reduction Off: To compare the advantage of the special noise reduction feature the tests will be done additionally with the deactivated feature.
  Feature for noise reduction (on): The noise reduction feature shall support the hearing aid user in noisy situations and shall reduce the listening effort.
  Feature for noise reduction (off): To show the advantage of the noise reduction feature there is a comparison without the feature necessary.
Arm/Group | Noise Reduction on | Noise Reduction Off
Number analyzed (Participants) | 8 | 8
SNR (dB) | -2.276 [-4.91 to 0.358] | -0.917 [-3.55 to 1.717]

2. Secondary Outcome: Subjective Ratings of Speech and Music Samples (Part1: Sound Quality)
Description: The secondary Outcome measure of this study contains 2 parts. This first part reported here was the evaluation of the sound quality. A comparison was made between speech and music audio excerpts either with or without gain being increased by the feedback manager.
  Subjective ratings of sound quality were made under both of these conditions for one speech and one music sample, using the following scale: Bad (1) - Poor (2) - Fair (3) - Good (4) - Excellent (5).
  Results were analyzed separately for the speech and music samples.
Time Frame: 4 weeks
Population: The test was done by 9 participants, but just the results of 8 participants could be used for the analysis.
  This is because technical limitations meant it was not possible to perform the test under both experimental conditions for one participant.
Measure: Median (Standard Deviation); unit: score on a scale
Groups:
- Evaluation of Sound Quality Without Increasing Gain: All participants had to evaluate the sound quality with the standard fitting of the feedback manager.
- Evaluation of Sound Quality With Increasing Gain: All participants had to evaluate the sound quality with additional gain, enabled by the feedback manager.
Arm/Group | Evaluation of Sound Quality Without Increasing Gain | Evaluation of Sound Quality With Increasing Gain
Number analyzed (Participants) | 8 | 8
score on a scale
  Speech sample | 4 (0.99) | 4 (1.16)
  Music sample | 3.5 (1.49) | 4 (1.07)

3. Secondary Outcome: Measure of Detection Threshold (in dB) for Soft Sounds
Description: This outcome measure evaluated the ability to detect sounds in a quiet environment.
  A comparison was made between the feature under investigation being activated and deactivated.
  Participants were asked to change the level of a speech sample until they were just able to detect it.
  The ability will be measured by a detection threshold (in dB).
Time Frame: 2 weeks
Measure: Median (Standard Deviation); unit: dB
Groups:
- Feature for Soft Noise on: A threshold was measured with activated feature.
- Feature for Soft Noise Off: A threshold was measured with deactivated feature.
Arm/Group | Feature for Soft Noise on | Feature for Soft Noise Off
Number analyzed (Participants) | 10 | 10
dB | 36.62 (8.1) | 38.21 (9.33)

4. Secondary Outcome: Subjective Ratings of Speech and Music Samples (Part 2: Artefact Perception)
Description: The second part of this secondary Outcome measure was the evaluation of audible artefacts either with or without the available gain being increased by the feedback manager.
  The outcome was measured as a binary response (artefacts audible/ not audible). Participants had to indicate whether artefacts were audible under both of these conditions.
  The number of positive ratings (artefacts were audible) was counted.
Time Frame: 2 week
Population: 9 participants completed this study period, but just the results of 8 participants could be used.
  This was because technical issues limited the reliability of the measures made for one participant.
  N.B. this test was independent from the other tests in the study. Therefore the results are not influenced by other test periods. The number of people included in the analysis described here relates only to this test.
Measure: Count of Participants; unit: Participants
Groups:
- Feedback Management Off: The participants shall evaluate if there are artefacts audible without additional gain, while hearing a recorded conversation
- Feedback Management on: The participants shall evaluate if there are artefacts audible with with additional gain, while hearing a recorded conversation
Arm/Group | Feedback Management Off | Feedback Management on
Number analyzed (Participants) | 8 | 8
Participants
  speech sample | 2 | 1
  music sample | 1 | 1

ADVERSE EVENTS:
Time Frame: 3.5 month
Groups:
- Events During the Test Period: During the test period no Adverse Events, serious adverse events or other events occured.
- Events Prior to Test Period (After Screening Appointment and Signed Informed Consent Form): The adverse events of this study were not related to the investigational device or to a test of the study.
  Therefore we report the adverse events in one group instead of each individual condition.
  The occurred events were prior to a test / study appointment. The adverse events occurred after the screening appointment, but before any intervention. Therefore the adverse events cannot be attributed to any single study condition. As such we report adverse events here simply for the entire study cohort.
Arm/Group | Events During the Test Period | Events Prior to Test Period (After Screening Appointment and Signed Informed Consent Form)
All-Cause Mortality (participants affected / at risk) | 0/9 | 0/9
Serious Adverse Events (participants affected / at risk) | 0/9 | 0/9
Other Adverse Events (participants affected / at risk) | 0/9 | 2/9
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Events During the Test Period (N=9) | Events Prior to Test Period (After Screening Appointment and Signed Informed Consent Form) (N=9)
Eye problem prior to first appointment (Eye disorders) | 0 (0) | 1 (1) — Prior to the first appointment, the participant informed that the first appointment is not possible, due to problems with the retina. This event was prior to the first study appointment and is not related to the study devices or study test procedure.
Ear infection (Infections and infestations) | 0 (0) | 1 (1) — In the first appointment the investigator noted an infection of the ear channel and canceled the appointment. No test was done and no device was placed on the ear at this time. The doctor confirmed that the participant is able to continue the study.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-12-17): https://cdn.clinicaltrials.gov/large-docs/73/NCT04723173/Prot_SAP_000.pdf